CLINICAL TRIAL: NCT03264014
Title: An Observational Pilot sTudy to Assess the Feasibility of Combining Data From Patient Registries in Countries With Developing Health Care Systems to EvaluaTe Haemophilia Management
Brief Title: Combining Registry Data in Haemophilia: TARGET H
Acronym: TARGET-H
Status: Completed | Type: Observational
Sponsor: University of Pretoria (Other)
Collaborators: Novo Nordisk A/S (Industry); Medical Research Council, South Africa (Other)
Responsible Party: Principal Investigator, Joachim Potgieter, Dr., University of Pretoria
Other Study IDs: UP TARGET H
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Haemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an investigator-initiated, multinational, retrospective, non-interventional pilot study conducted in five haemophilia treatment centres from different geographical regions that maintain a local (Algeria, Malaysia) or national (India, Iran, South Africa) haemophilia registry. Data from a randomly selected sample of patients from national or local registries are anonymously collated and analysed.The aims are to determine the feasibility of combining data from national and local registries in countries with developing healthcare systems and to assess how existing registries implemented current recommendations for data collection in terms of available fields and their completion.

DETAILED DESCRIPTION:
The study is conducted in five haemophilia treatment centres (HTCs) from different geographical regions (Algeria, India, Iran, Malaysia and South Africa) that maintain a local or national haemophilia registry. Data will be collected from 20 randomly selected, active patient records from each participating registry/country. In countries with national registries, data from local registries will not be permitted for inclusion to allow adequate assessment of the possibility of registry harmonisation across various regions. Participating centres will report data as available in the data source without seeking additional information to fill source data gaps at the time of data collection. In addition, each investigator will complete a basic questionnaire on feasibility parameters to confirm the source and accuracy of the data, as well as challenges experienced during data collection. Analysed parameters will be grouped into three categories: sociodemographic, disease, and treatment and disease outcome parameters. Feasibility assessment will be performed for all study variables and the percentage availability of each study variable recorded in the participating registries wii be determined, as well as the proportion of missing data for existing variables.

ELIGIBILITY:
Inclusion Criteria:

* male
* diagnosis of haemophilia A or B
* with or without inhibitors
* no other inherited bleeding disorder
* active patient record
* willing and able to provide written consent

Exclusion Criteria:

- unwilling or unable to provide written consent

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Registry records of 100 randomly selected haemophilia patients
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Haemophilia registry data | May to September 2015
  sosiodemographic parameters, disease parameters and treatment and disease outcome parameters